CLINICAL TRIAL: NCT02835443
Title: Electrical Stimulation of the Dentate Nucleus Area (EDEN) for Improvement of Upper Extremity Hemiparesis Due to Ischemic Stroke: A Safety and Feasibility Study
Brief Title: Electrical Stimulation of the Dentate Nucleus for Upper Extremity Hemiparesis Due to Ischemic Stroke
Acronym: EDEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enspire DBS Therapy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REDD 0002
Record Dates: First submitted 2016-07-07; First posted 2016-07-18 (Estimated); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Stroke
Keywords: Ischemic Stroke; Deep Brain Stimulation; DBS; Physical Therapy; Rehab; Brain Stimulation
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Electrical Stimulation (Experimental): This is a single arm study and all subjects will receive electrical stimulation.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Electrical stimulation of the dentate nucleus area of the cerebellum.

SUMMARY:
This clinical trial will evaluate if Deep Brain Stimulation (DBS) is safe for the treatment of stroke and will help understand if DBS improves motor recovery for patients who continue to have significant impairment.

DETAILED DESCRIPTION:
The proposed study is a safety and feasibility study intended to provide preliminary data to design a future pilot study. The objective of this study is to document the safety and patient outcomes of electrical stimulation of the dentate nucleus area for the management of chronic, moderate to severe upper extremity hemiparesis due to ischemic stroke.

ELIGIBILITY:
Key Inclusion Criteria:

* One-time stroke that occurred 1-3 years ago (i.e. index stroke 12-36 months)
* Stroke due to a blocked blood vessel (i.e. unilateral MCA stroke)
* Moderate to severe weakness in one arm (i.e. unilateral upper-extremity hemiparesis)

Key Exclusion Criteria:

* Seizures since time of stroke (i.e. seizures or seizure disorder)
* Unable to have an MRI (i.e. contraindicated for MRI)

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2023-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre Machado, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baker KB, Plow EB, Nagel S, Rosenfeldt AB, Gopalakrishnan R, Clark C, Wyant A, Schroedel M, Ozinga J 4th, Davidson S, Hogue O, Floden D, Chen J, Ford PJ, Sankary L, Huang X, Cunningham DA, DiFilippo FP, Hu B, Jones SE, Bethoux F, Wolf SL, Chae J, Machado AG. Cerebellar deep brain stimulation for chronic post-stroke motor rehabilitation: a phase I trial. Nat Med. 2023 Sep;29(9):2366-2374. doi: 10.1038/s41591-023-02507-0. Epub 2023 Aug 14. PMID 37580534

RESULTS

PARTICIPANT FLOW:
Groups:
- DBS+Rehab: This was a single-arm study, and all subjects received Deep Brain Stimulation (DBS) of the dentate nucleus area of the cerebellum plus rehab (DBS+Rehab)
Period: Overall Study
Arm/Group | DBS+Rehab
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DBS+Rehab
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Incidence of study-related serious adverse events
Time Frame: 18 Months
Measure: Number; unit: study-related, serious adverse events
Groups:
- DBS+Rehab: This was a single-arm study, and all subjects received Deep Brain Stimulation (DBS) of the dentate nucleus plus rehabilitation therapy (DBS+Rehab).
Arm/Group | DBS+Rehab
Number analyzed (Participants) | 12
study-related, serious adverse events | 0

ADVERSE EVENTS:
Time Frame: 18 Months
Arm/Group | DBS+Rehab
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBS+Rehab (N=12)
Low potassium / hypokalemia (Non Study-Related) (Blood and lymphatic system disorders) | 1 (1) — The subject went to a nearby Emergency Department for nausea and vomiting and was admitted for Hypokalemia; per definition, hospitalization is reported as an SAE. The subject had a history of Hypokalemia.
OTHER ADVERSE EVENTS (reported when occurring in more than .10% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DBS+Rehab (N=12)
Post-anesthesia nausea (Surgical and medical procedures) | 3 — See published article for details of all AEs: Baker KB, et al. Cerebellar deep brain stimulation for chronic post-stroke motor rehabilitation: a phase I trial. Nature Medicine. 2023;10.1038. https://doi.org/10.1038/s41591-023-02507-0
Post-surgical incision pain/sensitivity or headache (Surgical and medical procedures) | 6
IPG site pain/redness (Surgical and medical procedures) | 2
Nausea and vomiting during DBS programming (Surgical and medical procedures) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-12-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT02835443/Prot_000.pdf